CLINICAL TRIAL: NCT05572528
Title: Lenvatinib Therapy in the Patients With High-risk Hepatocellular Carcinoma After LDLT
Brief Title: Lenvatinib Therapy in HCC Patients After LDLT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaoshiung Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMRPG8M0041
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Liver Transplantation; Hepatocellular Carcinoma
Keywords: Liver transplantation Transplantation; Hepatocellular carcinoma; recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
New guidelines have been successfully established to distinguish the patients who were suitable for LT. This is important for long-term recurrence free and overall survival rate. We stratified patients with PET diagnosis and fetal protein response to confirm if they were the high-risk group for HCC recurrence. According to our new guidelines, high-risk tumor biology and tumor necrosis have important indicators for improving overall survival. Response to topical therapy is associated with tumor biology and post-transplant recurrence risk. In addition, the challenge of LDLT to HCC is that tumors with a high risk of recurrence have a high rate of recurrence after liver transplantation, and there is no appropriate treatment to prevent HCC recurrence after transplantation in these patients. Using the advance proton therapy or yttrium 90 as a more aggressive down-staging therapy may contribute to change tumor behavior. It can be used to get a better treatment response and tumor necrosis before LDLT. As a result, it will improve recurrence-free survival and overall survival rate, especially in high-risk groups.

In addition, lenvatinib is approved for using in patients with advanced liver cancer because its overall survival rate is not less than sorafenib in clinical trials. A new generation of targeted therapies will be applied to adjuvant therapy after LDLT.

DETAILED DESCRIPTION:
The research is an open, randomized, single-center study. Patients with high-risk recurrence of hepatocellular carcinoma who underwent liver transplantation are included according to the criteria of admission. Patients enrolled in the study were randomly allocated in the lenvatinib group (30 patients) after stable condition. We will use retrospective data to be as the control group. Patients in the control group are given supportive treatment and regular follow-up. Patients in the lenvatinib group are given lenvatinib within 1-2 months after operation (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day) for two years. The baseline data of patients are collected before allocation. Serum and imaging examination are checked regularly every month to monitor the recurrence of hepatocellular carcinoma and the side effects of lenvatinib. The efficacy and safety of lenvatinib in patients of high-risk hepatocellular carcinoma are observed, and the clinicopathological factors affecting the efficacy of lenvatinib are analyzed. When side effects of lenvatinib occur, the dosage can be reduced according to the patients' condition until discontinuation. When tumor recurrence occurs, a multidisciplinary team will draw up specific treatment plans according to the patients' condition, including surgical resection, interventional therapy, radiofrequency therapy, radiotherapy and targeted therapy.

Patients Criteria

Inclusion Criteria:

Enroll criteria

1. Male or female patients aged 18 to 75.
2. Targeted therapy is acceptable within 1-2 months after liver transplantation.
3. Immunosuppressive regimen consists of calcineurin inhibitor, mycophenolate mofetil and sirolimus.
4. All male and female participants must take reliable contraceptive measures during the trial and within four weeks after the end of the trial.
5. The definition of high-risk patients:
6. The PET scan is positive before LDLT;
7. Tumors beyond USCF criteria
8. Poorly-differentiated tumor;
9. The patients who has poor AFP response (under 15%)or AFPabove 400 ng/ml after LRT after conventional LRT (RFA, PEI or TACE)

Exclusion Criteria:

1. Life expectancy is less than 3 months
2. Patients are with other malignant tumors simultaneously.
3. Patients are anaphylaxis to the inactive ingredients of lenvatinib or drugs.
4. Pregnant or lactating women (Female participants need pregnancy test within 7 days before treatment).
5. Preoperative history of severe cardiovascular disease: congestive heart failure above NYHA grade 2; active coronary heart disease (myocardial infarction occurred within 6 months before entry into the study); severe arrhythmia requiring antiarrhythmic treatment (allowable use of beta-blockers or digoxin); uncontrolled hypertension.
6. History of HIV infection.
7. Severe clinical active infections (> NCI-CTCAE version 3.0).
8. Epilepsy patients requires medication (e.g. steroids or antiepileptic drugs).
9. Patients with kidney diseases requires renal dialysis.
10. Drug abuse, medical symptoms, mental illness or social status that may interfere with participants' participation in research or evaluation of research results.
11. Patients who could not swallow oral drugs, such as those with severe upper gastrointestinal obstruction and need gastric tube feeding.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 to 75.
* Targeted therapy is acceptable within 1-2 months after liver transplantation.
* Immunosuppressive regimen consists of calcineurin inhibitor, mycophenolate mofetil and sirolimus.
* All male and female participants must take reliable contraceptive measures during the trial and within four weeks after the end of the trial.
* The definition of high-risk patients:
* The PET scan is positive before LDLT;
* Tumors beyond USCF criteria
* Poorly-differentiated tumor;
* The patients who has poor AFP response (<15%)or AFP>400 ng/ml after LRT after conventional LRT (RFA、PEI or TACE)

Exclusion Criteria:

* Life expectancy is less than 3 months
* Patients are with other malignant tumors simultaneously.
* Patients are anaphylaxis to the inactive ingredients of lenvatinib or drugs.
* Pregnant or lactating women (Female participants need pregnancy test within 7 days before treatment).
* Preoperative history of severe cardiovascular disease: congestive heart failure > NYHA grade 2; active coronary heart disease (myocardial infarction occurred within 6 months before entry into the study); severe arrhythmia requiring antiarrhythmic treatment (allowable use of beta-blockers or digoxin); uncontrolled hypertension.
* History of HIV infection.
* Severe clinical active infections (> NCI-CTCAE version 3.0).
* Epilepsy patients requires medication (e.g. steroids or antiepileptic drugs).
* Patients with kidney diseases requires renal dialysis.
* Drug abuse, medical symptoms, mental illness or social status that may interfere with participants' participation in research or evaluation of research results.
* Patients who could not swallow oral drugs, such as those with severe upper gastrointestinal obstruction and need gastric tube feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Although transplant consensus recommends surveillance for recurrent HCC after LT, its early diagnosis after LT has not been associated with improved survival or reduced cancer-related mortality. This scenario is probably related to the lack of curative treatments in these patients.
  Moreover, recurrence occurring during the first 2 years after transplant has been associated with even worse post-recurrence survival (PRS). Early recurrences may represent an aggressive HCC with worse biological behavior after transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The recurrence rate after LDLT in high risk patients | follow-up to two years
  High risk of recurrence usually occured in two years

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Cheng Gang, Kaohsiung City, Taiwan